CLINICAL TRIAL: NCT00003464
Title: Phase II Treatment of Adults With Newly Diagnosed Primary Malignant Glioblastoma Multiforme With Temodal
Brief Title: Temozolomide in Treating Adults With Newly Diagnosed Primary Malignant Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Henry Friedman, MD, Duke UMC
Purpose: Treatment
Other Study IDs: 1171; DUMC-1171-01-6R4; DUMC-1016-97-7; DUMC-1056-98-7R1; DUMC-1058-98-7R1; DUMC-1171-00-6R3; DUMC-1231-99-7R2; DUMC-97081; NCI-G98-1465; CDR0000066498 (Other: NCI)
Record Dates: First submitted 1999-11-01; First posted 2003-08-20 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2009-10

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — Temozolomide; Radiotherapy

INTERVENTIONS:
Drug: temozolomide
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of temozolomide in treating adults with newly diagnosed primary malignant glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor activity of temozolomide in adults with newly diagnosed glioblastoma multiforme.
* Define the relationship between tumor O6-alkylguanine-DNA alkyltransferase activity and tumor response in these patients.
* Define the relationship between tumor DNA mismatch repair activity and tumor response to temozolomide.

OUTLINE: Patients receive temozolomide orally once daily on days 1-5. Treatment courses are repeated every 28 days. In the absence of disease progression and toxicity, patients receive up to 4 courses of treatment prior to radiation therapy. After radiation therapy, patients demonstrating partial or complete response may receive an additional 12 courses of treatment.

Patients are followed every 8-12 weeks for 2 years.

PROJECTED ACCRUAL: This study will accrue 50 patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven, newly diagnosed, supratentorial malignant glioblastoma multiforme not requiring immediate radiation therapy
* At least 1 bidimensionally measurable lesion

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* Greater than 12 weeks

Hematopoietic:

* Absolute neutrophil count at least 1500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic:

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* SGOT and SGPT less than 2.5 times ULN
* Alkaline phosphatase less than 2 times ULN

Renal:

* BUN less than 1.5 times ULN
* Creatinine less than 1.5 times ULN

Other:

* Must be neurologically stable
* No systemic disease
* No acute infection requiring intravenous antibiotics
* No frequent vomiting
* No other medical condition that would interfere with oral medication intake such as partial bowel obstruction
* No prior or concurrent malignancies except:

  * Surgically cured carcinoma in situ of the cervix
  * Basal or squamous cell carcinoma of the skin
* HIV negative
* No AIDS-related illness
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior biologic therapy
* No concurrent biologic therapy (growth factors or erythropoietin)

Chemotherapy:

* No prior chemotherapy
* No other concurrent chemotherapy

Endocrine therapy:

* Concurrent steroid allowed (must be on stable dose for at least 1 week prior to study)

Radiotherapy:

* No prior radiation therapy
* No prior interstitial brachytherapy
* No prior radiosurgery to the brain
* Not requiring immediate radiation therapy
* No concurrent radiotherapy

Surgery:

* Recovered from any effects of prior surgery
* At least 2 weeks since prior surgical resection

Other:

* No other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 1997-09; Study Completion 2003-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry S. Friedman, MD, Study Chair — Duke University
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States